CLINICAL TRIAL: NCT02862496
Title: Urine N-telopeptide, Serum Vit D, Parathormone and Calcium Levels in Hyperemesis Gravidarum
Brief Title: Bone Health in Hyperemesis Gravidarum
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Kayseri Education and Research Hospital (Other Government)
Responsible Party: Principal Investigator, Erdem Sahin, Principal Investigator, Kayseri Education and Research Hospital
Other Study IDs: 2016/345
Record Dates: First submitted 2016-07-21; First posted 2016-08-11 (Estimated); Last update posted 2016-08-11 (Estimated); Status verified 2016-08

CONDITIONS: Hyperemesis Gravidarum
Keywords: Hyperemesis Gravidarum; Bone Health; Urine N-telopeptide; Serum calcium; Serum parathormone; Serum vit D
MeSH Terms: conditions — Hyperemesis Gravidarum

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 9 Months

GROUPS / COHORTS (2):
- hyperemesis gravidarum: hyperemesis gravidarum group consisting of 30 pregnant women between 7-20 weeks of gestation with diagnosed hyperemesis gravidarum.
- Control group: control group consisting of 30 health pregnant women between 7-20 weeks of gestation with excluded hyperemesis gravidarum.

SUMMARY:
The purpose of the study is to determine whether maternal bone resorption would be seen in Hyperemesis Gravidarum and could be detected in early period using serum vitamin D levels, serum calcium (Ca) levels, serum parathormone (PTH) levels and urine N- telopeptide levels in the patients with Hyperemesis Gravidarum.

ELIGIBILITY:
Inclusion Criteria:

* Between 7. and 20. weeks of gestation pregnant women in both groups
* İn hyperemesis group; 5% weight loss with regard to pre-gestation vomiting more than 3 times 3-5 % weight loss with ketonuria.

Exclusion Criteria:

* Other pathologies that cause nausea and vomiting in pregnancy gastroenteritis gastroparesis gall duct diseases hepatitis peptic ulcers appendicitis pyelonephritis ovarian torsion urinary tract stones diabetic ketoacidosis hyperthyroidism hyperparathyroidism migraine pseudo tumor cerebra vestibular diseases
* Additionally some situations causing to rise of Ntx levels osteoporosis paget disease bone tumors
* Furthermore some of conditions resulted in pre-menopausal osteoporosis or decreasing in Bone Mineral Density Malignancy Smoking Celiac Disease Depression Inflammatory Bowel Disease Pre-gestational Diabetes Chronic Kidney or Liver Disease Drug Use such as steroids, anticonvulsants, antiepileptic, heparin or low molecular weight heparin

Ages: 18 Years to 35 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: The study population was consisted of 2 groups and included pregnant women in between 7. and 20. weeks of gestation for both groups. The normal pregnancy group was consisted of 30 healthy pregnant women whom excluded hyperemesis gravidarum (HG), the HG group was consisted of 30 pregnant women with diagnosed HG.
Sampling Method: Non-Probability Sample
Enrollment: 60 (Estimated)
Dates: Start 2016-06; Primary Completion 2016-10 (Estimated); Study Completion 2016-10 (Estimated)

PRIMARY OUTCOMES:
Urine N- telopeptide levels in Pregnant Women with Hyperemesis Gravidarum | 4 months
Serum Vitamin D Levels in Pregnant Women with Hyperemesis Gravidarum | 4 months
Serum Calcium Levels in Pregnant Women with Hyperemesis Gravidarum | 4 months
Serum Parathormone Levels in Pregnant Women with Hyperemesis Gravidarum | 4 months

CONTACTS AND LOCATIONS:
Overall Officials: Erdem SAHİN, Study Director — Kayseri Training and Research Hospital
Locations (1):
- Kayseri Training and Research Hospital, Kayseri, Turkey (Türkiye)

REFERENCES:
- [Background] Bailit JL. Hyperemesis gravidarium: Epidemiologic findings from a large cohort. Am J Obstet Gynecol. 2005 Sep;193(3 Pt 1):811-4. doi: 10.1016/j.ajog.2005.02.132. PMID 16150279
- [Background] Minami H, Furuhashi M, Minami K, Miyazaki K, Yoshida K, Ishikawa K. Fetal intraventricular bleeding possibly due to maternal vitamin K deficiency. Fetal Diagn Ther. 2008;24(4):357-60. doi: 10.1159/000163078. Epub 2008 Oct 16. PMID 18931500
- [Background] Yahia M, Najeh H, Zied H, Khalaf M, Salah AM, Sofienne BM, Laidi B, Hamed J, Hayenne M. Wernicke's encephalopathy: A rare complication of hyperemesis gravidarum. Anaesth Crit Care Pain Med. 2015 Jun;34(3):173-7. doi: 10.1016/j.accpm.2014.09.005. Epub 2015 May 21. No abstract available. PMID 26004883
- [Background] Practice Bulletin No. 153: Nausea and Vomiting of Pregnancy. Obstet Gynecol. 2015 Sep;126(3):e12-e24. doi: 10.1097/AOG.0000000000001048. PMID 26287788
- [Background] Hanson DA, Weis MA, Bollen AM, Maslan SL, Singer FR, Eyre DR. A specific immunoassay for monitoring human bone resorption: quantitation of type I collagen cross-linked N-telopeptides in urine. J Bone Miner Res. 1992 Nov;7(11):1251-8. doi: 10.1002/jbmr.5650071119. PMID 1466251
- [Background] Hlaing TT, Compston JE. Biochemical markers of bone turnover - uses and limitations. Ann Clin Biochem. 2014 Mar;51(Pt 2):189-202. doi: 10.1177/0004563213515190. Epub 2014 Jan 7. PMID 24399365
- [Background] Sanz-Salvador L, Garcia-Perez MA, Tarin JJ, Cano A. Bone metabolic changes during pregnancy: a period of vulnerability to osteoporosis and fracture. Eur J Endocrinol. 2015 Feb;172(2):R53-65. doi: 10.1530/EJE-14-0424. Epub 2014 Sep 10. PMID 25209679
- [Derived] Sahin E, Madendag Y, Eraslan Sahin M, Tayyar AT, Col Madendag I, Gozukucuk M, Karakukcu C, Acmaz G, Muderris II. Maternal type 1collagen N-terminal telopeptide levels in severe hyperemesis gravidarum. BMC Pregnancy Childbirth. 2018 Dec 20;18(1):502. doi: 10.1186/s12884-018-2149-7. PMID 30572827